CLINICAL TRIAL: NCT01082900
Title: Prophylactic CPAP/PEEP in Delivery Room (DR) Resuscitation, Effects on Natriuretic Peptide in the Prevention of Transient Tachypnea of Newborn (TTN): A Randomized Controlled Trial
Brief Title: Prophylactic Continuous Positive Airway Pressure (CPAP) in Delivery Room, in the Prevention of Transient Tachypnea of Newborn (TTN): A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Hospital Queens (Other)
Responsible Party: Principal Investigator, pinchi srinivasan, MD, New York Hospital Queens
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 5720108
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Transient Tachypnea
Keywords: Transient Tachypnea of the Newborn; Elective Cesarean section; Late preterm; CPAP; Delivery Room
MeSH Terms: conditions — Transient Tachypnea of the Newborn

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylactic CPAP intervention (Experimental): Babies will receive prophylactic administration of CPAP (5 cm of H2O) in the DR via T piece (Neopuff)
  Interventions: Other: Prophylactic CPAP Administration
- No Intervention (Active Comparator): Provision of standard care in the Delivery Room
  Interventions: Other: Prophylactic CPAP Administration

INTERVENTIONS:
Other: Prophylactic CPAP Administration — EXPERIMENTAL GROUP: Babies will receive prophylactic administration of CPAP (5 cm of H2O) in the Delivery Room via T piece (Neopuff)
  CONTROL GROUP: Provision of standard care in the Delivery Room

SUMMARY:
Transient Tachypnea of the Newborn (TTN) is a disorder of delayed clearance of lung liquid and a common cause of admission of full term infants and late pre term infants (34 to 36 weeks) to Neonatal Intensive Care Units (NICU). Both late preterm gestational age at delivery, and mode of delivery are considered risk factors for TTN. The investigators hypothesize that CPAP administered prophylactically in the Delivery Room via a T piece based infant resuscitator Neopuff, to neonates at increased risk for TTN, would decrease the incidence of TTN and thus decrease the need for hospitalization in the NICU. This is a pilot study to evaluate the prophylactic administration of CPAP in the Delivery Room towards prevention of TTN and it's effects on natriuretic peptides.The study will be conducted as a randomized control trial after obtaining informed consents from the parents of eligible infants. Infants will be randomized to receive either experimental treatment (prophylactic CPAP) or standardized care.

ELIGIBILITY:
Inclusion Criteria:

* Babies born to mothers via elective CS: elective CS defined as planned CS in the absence of Labor.
* Late preterm infants (34 1/7 to 36 6/7 weeks gestational age)

Exclusion Criteria:

* Presence of any of the risk factors for neonatal sepsis such as Prolonged Rupture of Membranes for ≥18 hours (PROM), maternal fever, maternal chorioamnionitis or positive maternal GBS colonization
* Need for use of PPV for perinatal depression or other indications
* Presence of any of the following

  * congenital malformations (diagnosed prenatally)
  * chromosomal anomalies (diagnosed prenatally)
  * congenital heart disease diagnosed by fetal echocardiography.

Ages: 2 Minutes to 30 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2009-11; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Measure of incidence of TTN | 24 hours
Need for admissions to NICU secondary to TTN | 24 hours

SECONDARY OUTCOMES:
levels of plasma brain natriuretic peptide compared | 24 hours
  * Duration of tachypnea
  * Duration of oxygen therapy
  * Length of hospital (NICU) stay

CONTACTS AND LOCATIONS:
Overall Officials: Pinchi Srinivasan, MD, Principal Investigator — New York Hospital Queens
Locations (1):
- New York Hospital Queens, Flushing, New York, United States